CLINICAL TRIAL: NCT03997994
Title: Drug-Coated Balloon for the Treatment of Symptomatic Chronic Benign Biliary Stricture
Brief Title: DIGEST I Drug Coated Balloon for Biliary Stricture
Acronym: DIGEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GIE Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR 2002
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Biliary Stricture; Biliary Anastomotic Stenosis; Biliary Obstruction; Biliary Disease
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental: DCB Treatment (Experimental): Stricture patients treated by DCB
  Interventions: Device: GIE Drug Coated Balloon

INTERVENTIONS:
Device: GIE Drug Coated Balloon — The GIE DCB is a balloon catheter coated with a proprietary coating containing the drug and carriers.

SUMMARY:
DIGEST I Pilot study is a feasibility study for evaluating the safety and efficacy of DCBs.

DETAILED DESCRIPTION:
The study is designed to determine the safety and effectiveness of drug coated balloon (DCB) treatments on biliary tract stricture.

Up to 15 subjects are planned to be enrolled and treated with the study device at up to 5 clinical sites outside of US. Subjects will be followed up post-treatment to one year and then annually for up to 5 years. The annual follow up after the first year is optional.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years.
2. Benign biliary stricture with postoperative injury or PSC or anastomotic-stricture; and indicated for ERCP procedure.
3. Restenosis after plain balloon dilation with at least 2 previous balloon dilation sessions and recurrence of biliary obstructive symptoms/signs or being managed with implantable prosthetics (e.g. plastic stents).
4. Greater than 40% stenosis of the biliary tract via ERCP.
5. Total serum bilirubin >2 mg/dL. Alkaline phosphatase level >3 times higher than normal level. *Note: This IC is waved if the patient is being managed with implantable prosthetics.
6. Type I, II, III and IV Benign biliary duct strictures. Dominant stricture being accessible by balloon catheter.
7. Stricture length <4 cm.
8. Not currently listed for liver transplantation.
9. Voluntary participation and provided written informed consent.

Exclusion Criteria:

1. Pregnancy or breastfeeding or plan to get pregnant in next 12 months.
2. Benign biliary strictures caused by pancreatic pseudocyst compression.
3. Malignant biliary obstruction.
4. Biliary obstruction associated with an attack of acute pancreatitis.
5. Inability to pass guidewire across stricture.
6. Subjects with cholangitis or bile leak or duct fistula.
7. Contraindication for Endoscopic Retrograde Cholangiopancreatography (ERCP) or anesthesia or deep sedation or MRI.
8. Subject with an internal/external biliary drainage catheter.
9. Subjects with surgically altered gastro/duodenal/jejunal anatomy (e.g. Roux-Y-loop, choledochojejunostomy).
10. Subject with symptomatic duodenal stenosis (with gastric stasis)
11. Active systemic infection.
12. Allergy to paclitaxel or any components of the delivery system.
13. Currently undergoing required thoracic or abdominal cavity radiation therapy.
14. Has life expectancy <12 months.
15. Unwilling or unable to comply with the follow-up study requirements.
16. Lacking capacity to provide informed consent.
17. Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety.
18. Currently participation in another pre-market drug or medical device clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-12 (Actual); Primary Completion 2024-03-21 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
Incident of serious balloon dilation-related complications | 30 days
  No serious procedure-related complications, including perforation, bleeding requiring invasive intervention or transfusion, cholangitis, pancreatitis, etc.
Freedom from Biliary Stricture Re-intervention | 12 months
  Biliary stricture re-intervention rate

SECONDARY OUTCOMES:
Change in Liver Function | Baseline, 7 days, 30 days, 3 months, 6 months, 12 months and 24 months
  . Liver function tests include total and direct bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT)
Change in Existing Biliary Obstructive Symptoms | Baseline, 30 days, 3 months, 6 months, 12 months and 24 months
  The common biliary obstructive symptoms are right upper quadrant pain (survey), fever/chills (cholangitis), jaundice, itching, dark urine, pale stools, nausea/vomiting, weight loss
Biliary Stricture Diameter | Baseline, 6 months
  Stricture diameter will be assessed via endoscopic retrograde cholangiopancreatography (ERCP)
Time to the First Re-intervention | 12 months and 24 months
  The mean time to the first re-intervention (scheduled and unscheduled) will be assessed
Sustained Clinical Success (SCS) | 12 months and 24 months
  SCS defined as a period of at least 6 months with no need for further endoscopic intervention
Long Term Clinical Success (LTCS) | 12 months and 24 months
  LTCS, defined as no need for further endoscopic intervention for at least 24 months
Mean number of dilations | 12 months and 24 months
  Mean number of dilations required to achieve SCS and LTCS
Technical Success | 0 months
  Technical success is defined as successful insertion, dilatation of the target biliary stricture, and finally withdrawal of the device with no device malfunctions.

CONTACTS AND LOCATIONS:
Overall Officials: Bret T Petersen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Adventista Hospital, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: Undecided